CLINICAL TRIAL: NCT04521244
Title: Immediate Effects of Thrust Versus Non-thrust Lumbar Manipulation on Mobility and Springing Force Tolerance in Lumbar Hypomobility
Brief Title: Lumbar Manipulation in Lumbar Hypomobility
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC/00695 Saba Nawaz
Record Dates: First submitted 2020-08-18; First posted 2020-08-20 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Hypomotility; Lumbar Spine Instability
Keywords: Lumbar Mobilization; Hypo-mobility; Spinal or segmental stiffness; Lumbar Manipulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Thrust joint lumbar manipulation (Experimental): Thrust joint lumbar manipulation (Lumbar rotation manipulation) ,Moist Hot pack
  Interventions: Other: Thrust joint lumbar manipulation
- Lumbar mobilization (Active Comparator): Lumbar mobilization (Stretch rotation mobilization), Moist Hot pack
  Interventions: Other: Lumbar mobilization

INTERVENTIONS:
Other: Thrust joint lumbar manipulation — Moist Hot pack of 14/15' over lumbar region for 15 mins. Hydro collator Temperature according to standardized hot pack is 40-45οC.Bilateral Thrust Manipulation of Lumbar Spine from L1-L5 Baseline Algometer for springing force tolerance and Lumbar Inclinometry using dual inclinometer for lumbar flexion, extension and goniometer for lumbar side bending.These pre and post intervention values were mentioned in questionnaire. The participants were administered with thrust and non-thrust manipulation of the lumbar spine and data was collected again immediately after the interventions without any delay.
  Arms: Thrust joint lumbar manipulation
Other: Lumbar mobilization — Moist Hot pack of 14/15' from L1 where ribcage ends up to the region of gluteal folds for 15 mins. Non Thrust Manipulation for 30 seconds Using Kaltenborn grade 3 (Stretch rotation mobilization).Baseline Algometer for springing force tolerance and Lumbar Inclinometry using dual inclinometerfor lumbar flexion, extension and goniometer for lumbar side bending. These pre and post intervention values were mentioned in questionnaire. The participants were administered with thrust and non-thrust manipulation of the lumbar spine and data was collected again immediately after the interventions without any delay.
  Arms: Lumbar mobilization

SUMMARY:
The purpose of the study is to compare the immediate effects of thrust versus non-thrust lumbar manipulation in individuals with lumbar hypo-mobility on lumbar range of motion and springing force tolerance. A randomized control trial was conducted at Max Rehab and Physical Therapy Centre, Islamabad. The sample size was 18 calculated through open-epi tool but I recruited 60. The participants were divided into two interventional groups each having 30 participants. The study duration was six months. Sampling technique applied was Purposive sampling for recruitment and group randomization using flip coin method. Only 20 to 35 years participants with grade one or two hypo-mobility at lumbar region were included in the study. Tools used in this study are Goniometer, Inclinometers (lumbar Inclinometry using dual inclinometer method),Digital Algometer, Self structured Questionnaire. Data was collected before and immediately after the application of interventions. Data analyzed through SPSS version 23.

DETAILED DESCRIPTION:
A systematic and evidence based search of relevant literature was performed by utilizing PubMed and Google Scholar as search engines and the key words used were lumbar manipulation, hypo-mobility, spinal stiffness, non-thrust manipulation, lumbar mobilizations, segmentalstiffness.The purpose of the literature review is to find out the pre-existing literature regarding the Lumbar mobilizations and TJM interventions for Lumbar Hypomobility.

In 2019 a systematic review conducted by Aoyagi et al on effectiveness of spinal mobilization stated that there is a moderate to high quality evidence on Spinal mobilizations as effective intervention in low back pain as it decreases pain and improve Range of motion In 2019,a systematic review conducted by Hofstetter et al on Instrumented measurement of spinal stiffness stated that mechanical devices revealed excellent reliability tool to measure Spinal stiffness especially in prone position.

In 2019, a systematic review and meta-analysis conducted by a chi Ngai Lo et al on Spinal manipulation stated that HVLAT is highly effective as an treatment protocol then no intervention or sham manipulation because it improves muscle strength in healthy population

ELIGIBILITY:
Inclusion Criteria:

* Both Genders
* Participants having Lumbar flexion ≤ 30ᴼ
* Participants having lumbar extension ≤15ᴼ
* Participants having lumbar side bending ≤ 15ᴼ.
* Grade 1 & 2 hypo-mobility (Stanley Paris Grading System)
* Springing force tolerance measured through Pressure Algometry using Digital
* Algometer whose value can be taken in kg or lb.
* Checklist of Red Flags of TJM Lumbar Spine (Tumor, any bacterial or viral infection like Tuberculosis, UTI which is accompanying any neurological impairments i.e loss of sensations in extremities, Severe Rheumatoid Arthritis,Osteomalacia or Osteoporosis, cervical myelopathy, cord compression,cauda equina syndrome, Bowel and bladder changes, motor vehicle accident or fall, Muscle weakness or atrophy, any history of immunosuppression e.g. steroids, HIV, Abnormal Deep tendon reflexes, Headache, confusion, Abnormal and constant changes in pain pattern, Bilateral or Unilateral Sciatica.)

Exclusion Criteria:

* Participants having normomobility and hypermobility (according to Beighton Score, a score of 4 or more out of 9 indicates generalized hypermobility of the Joints).
* Participants having fracture and lumbar prolapsed intervertebral disc
* Participants having Spondylolisthesis, Lumbar Trauma, any musculoskeletal or cardiorespiratory disorders that affects lumbar spine mobility like (SI, Hip Joint, Thoracic Spine dysfunction)
* Participants who received any therapy for lumbar region past 3 days

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2019-11-05 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-11-09 (Actual)

PRIMARY OUTCOMES:
Stanley Paris Grading (Self-Structured Questionnaire and Screening Questionnaire) | On Day 1
  It is 0-6 PIVM Grading system for manual grading of Rotatoric Movement.From 0-2 grades considered as Hypo-mobility. Grade 1 is considerable decreased movement and grade 2 is slight decreased movement at the lumbar region.As per my inclusion criteria, participants with grade 1 & 2 hypo-mobility were included.On the basis of screening questionnaire, lumbar hypo-mobility was diagnosed by Stanley Paris grading system and after taking demographics in self-structured questionnaire, pre and post intervention values were mentioned in the Questionnaire.0 grade is no movement (ankylosis or fused) while 6 grade is complete instability.
ROM Lumbar spine ( Flexion) | On Day 1
  Participants having lumbar flexion ≤ 30° were recruited.Changes from the Baseline ROM (range of Motion) of Lumbar flexion was taken with the Help of Inclinometers. Standard normative value for lumbar range for flexion is 40-60°.
ROM Lumbar spine (Extension) | On Day 1
  Participants having lumbar extension ≤ 15° were recruited. Changes from the Baseline ROM (range of Motion) of Lumbar extension was taken with the Help of Inclinometers. Standard normative value for lumbar range of extension is 20-35°.
ROM Lumbar spine (Side Bending) | On Day 1
  Participants having side bending ≤ 15° were recruited.Changes from the Baseline ROM (range of Motion) of Lumbar side bending was taken with the Help of Goniometer. Standard normative value for lumbar range of side bending is 15-20°.

SECONDARY OUTCOMES:
Pressure Pain Threshold (PPT) | On Day 1
  Changes from Baseline Pressure Pain Threshold (PPT) were taken with the help of digital algometer.which measures springing force tolerance in kg or lb.

CONTACTS AND LOCATIONS:
Overall Officials: Lal Gul Khan, MScPT, Principal Investigator — Riphah International University
Locations (1):
- Max Health, Islamabad, Fedral, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Coulter ID, Crawford C, Hurwitz EL, Vernon H, Khorsan R, Suttorp Booth M, Herman PM. Manipulation and mobilization for treating chronic low back pain: a systematic review and meta-analysis. Spine J. 2018 May;18(5):866-879. doi: 10.1016/j.spinee.2018.01.013. Epub 2018 Jan 31. PMID 29371112
- [Background] Hurwitz EL, Randhawa K, Torres P, Yu H, Verville L, Hartvigsen J, Cote P, Haldeman S. The Global Spine Care Initiative: a systematic review of individual and community-based burden of spinal disorders in rural populations in low- and middle-income communities. Eur Spine J. 2018 Sep;27(Suppl 6):802-815. doi: 10.1007/s00586-017-5393-z. Epub 2017 Dec 27. PMID 29282539
- [Background] Hoy D, March L, Brooks P, Blyth F, Woolf A, Bain C, Williams G, Smith E, Vos T, Barendregt J, Murray C, Burstein R, Buchbinder R. The global burden of low back pain: estimates from the Global Burden of Disease 2010 study. Ann Rheum Dis. 2014 Jun;73(6):968-74. doi: 10.1136/annrheumdis-2013-204428. Epub 2014 Mar 24. PMID 24665116
- [Background] Olotu JE, Okon M. Prevalence of Low Back Pain in a Southern Nigerian Population.
- [Background] Yang K. Outpatient rehabilitation for a patient with chronic low back stiffness. 2019.
- [Background] Petersson M, Abbott A. Lumbar interspinous pressure pain threshold values for healthy young men and women and the effect of prolonged fully flexed lumbar sitting posture: An observational study. World J Orthop. 2020 Mar 18;11(3):158-166. doi: 10.5312/wjo.v11.i3.158. eCollection 2020 Mar 18. PMID 32280605
- [Background] Page I, Descarreaux M. Effects of spinal manipulative therapy biomechanical parameters on clinical and biomechanical outcomes of participants with chronic thoracic pain: a randomized controlled experimental trial. BMC Musculoskelet Disord. 2019 Jan 18;20(1):29. doi: 10.1186/s12891-019-2408-4. PMID 30658622
- [Background] Aoyagi K, Heller D, Hazlewood D, Sharma N, Dos Santos M. Is spinal mobilization effective for low back pain?: A systematic review. Complement Ther Clin Pract. 2019 Feb;34:51-63. doi: 10.1016/j.ctcp.2018.11.003. Epub 2018 Nov 5. No abstract available. PMID 30712746
- [Background] Hofstetter L, Hausler M, Wirth B, Swanenburg J. Instrumented Measurement of Spinal Stiffness: A Systematic Literature Review of Reliability. J Manipulative Physiol Ther. 2018 Oct;41(8):704-711. doi: 10.1016/j.jmpt.2018.03.002. Epub 2019 Jan 3. PMID 30612717
- [Background] Lo CN, Ng J, Au CK, Lim ECW. The Effectiveness of Spinal Manipulation in Increasing Muscle Strength in Healthy Individuals: A Systematic Review and Meta-Analysis. J Manipulative Physiol Ther. 2019 Feb;42(2):148-158. doi: 10.1016/j.jmpt.2018.10.003. PMID 31126523